CLINICAL TRIAL: NCT04967313
Title: A Randomized, Controlled Trial to Test Behavior Change Techniques (BCTs) to Improve Low Intensity Physical Activity in Older Adults
Brief Title: Behavior Change Techniques (BCTs) to Improve Low Intensity Physical Activity in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Karina Davidson, Senior Vice President, Research & Dean of Academic Affairs, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-1166; 1P30AG063786-01 (NIH)
Record Dates: First submitted 2021-07-02; First posted 2021-07-19 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Sedentary Behavior
Keywords: Physical Activity; Sedentary Behavior; Behavior Change; Behavior Change Techniques; Virtual; Personalized Trial; Personalized; Feasibility
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: The order of administration for the 4 Behavioral Change Techniques (BCTs) will be randomized by the study statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Change Techniques to Increase Walking (Experimental): Individuals will receive daily text messages with the goal of increasing daily walking by 2,000 more steps five days per week. Participants will be enrolled for a baseline period lasting two weeks where their average daily activity level will be assessed using a Fitbit device to generate an average daily step counts. Following completion of baseline, participants will receive daily text messages of behavior change techniques (BCTs) for eight weeks. The four BCTs utilized in this study are: goal setting, action planning, self-monitoring of behavior, and feedback on behavior. Each BCT will be delivered to participants daily for a two-week block. Four blocks (one BCT per block) will be delivered to the participant. The order in which the BCT interventions are presented to participants will be randomized by the study statistician. The goal of the BCT text messages will be to encourage walking behavior.
  Interventions: Behavioral: Behavioral Change Techniques

INTERVENTIONS:
Behavioral: Behavioral Change Techniques — Four behavioral changes techniques (BCTs) will be administered to participants in random order. The BCTs are defined as follows:
  1. Goal setting: set or agree on a goal defined in terms of behavior to be achieved. Example: Set the goal of walking 2,000 steps more per day.
  2. Action planning: prompt detailed planning of performance of behavior (must include a setting [walking to the mailbox], frequency, duration, and intensity. Example: Develop a plan to walk today.
  3. Self-Monitoring of behavior: establish a method for person to monitor and record their number of steps based on their Fitbit. Example: Did you check your Fitbit and record daily total number of steps?
  4. Feedback on behavior: Monitor and provide informative or evaluative feedback on performance of the behavior (e.g. form, frequency, duration, intensity). Example: You walked 6,000 steps today. This is 1,000 steps above your baseline.

SUMMARY:
The purpose of this pilot study is to determine the feasibility of using personalized trial methods in a virtual research study with Northwell employees aged 45-75 years old to increase low-intensity walking by 2,000 steps per day/5 days per week using four behavior change techniques (BCTs), provided in random order, and shown to have been effective in changing physical activity. The study will include a two-week baseline period during which levels of physical activity and adherence to the trial protocol will be evaluated. Individuals meeting adherence criteria will be randomized to the eight-week BCT intervention.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility of using personalized trial methods in a virtual research study with Northwell employees aged 45-75 years old to increase low-intensity walking by 2,000 steps per day/five days per week using four behavior change techniques (BCTs), provided in random order, and shown to have been effective in changing physical activity. This pilot will help determine if a personalized, virtual trial design can have widespread use in future research and clinical practice. The investigators will randomize 60 participants. Participants will complete a two-week baseline period during which they will be asked to wear a Fitbit device all day and night, even while they are sleeping, and to acknowledge receipt of a daily text message that is not an activity prompt. Baseline participants will be instructed to sync their Fitbit device by opening the Fitbit app on their phone at least every two days. After completion of the baseline period, a clinical research coordinator will review individual adherence to Fitbit wear and to survey responses. Adherence to Fitbit wear will be defined as recorded activity of greater than 10 hours a day. Text message adherence will be defined as responding to a given text message. Baseline participants that do not achieve at least 80% adherence of Fitbit wear and text responsiveness during the two weeks of the baseline period will be withdrawn from the study. Those that maintain at least 80% adherence will be randomized to one of their selected behavior change techniques to begin their pilot personalized trial. Participants who are randomized to receive intervention sequences will receive email confirmation including their protocol timeline. Enrollment will continue until up to 60 participants have been randomized. Individuals in the intervention period will receive four BCTs: goal setting, action planning, self-monitoring of behavior, and feedback on behavior. BCTs will be delivered individually to participants over the course of eight weeks in four two-week blocks. The order of BCT administration will be randomized by the study statistician. Participants may receive additional text messages to those outlined above with important reminders to sync their data as needed. Upon completion, participants in the personalized trials phase will receive an individual report that demonstrates their walking responses in relation to their selected BCTs. After receiving the report, clinical research coordinators will contact participants to respond to questions and to obtain feedback about their personalized trials experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 75 years old of age
* Fluent in English
* Employed in the Northwell Health system
* Community-dwelling
* Report they are in good general health, walk regularly and have never been informed by a clinician that it was not advisable/safe to participate in a low-intensity walking program
* Owns and can regularly access a smartphone capable of receiving text messages
* Owns and can regularly access an e-mail account

Exclusion Criteria:

* < 45 years old or > 75 years old
* Unable to speak/comprehend English
* Not employed in Northwell Health system
* Have self-reported poor health, limited mobility and/or have been advised by a clinician not to increase their low-intensity walking
* Pregnancy
* Previous diagnosis of a serious mental health condition or psychiatric disorder, such as bipolar disorder

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Center for Personalized Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary. Pooling personalized trials together is a more efficient approach for deriving population-level estimates than conventional randomized controlled trials.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

REFERENCES:
- [Derived] Friel CP, Robles PL, Butler M, Pahlevan-Ibrekic C, Duer-Hefele J, Vicari F, Chandereng T, Cheung K, Suls J, Davidson KW. Testing Behavior Change Techniques to Increase Physical Activity in Middle-Aged and Older Adults: Protocol for a Randomized Personalized Trial Series. JMIR Res Protoc. 2023 Jun 14;12:e43418. doi: 10.2196/43418. PMID 37314839

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were consented and entered a 2-week baseline period prior to beginning the intervention. Participants who were not compliant with trial requirements during baseline did not continue to receive the intervention. Data were collected for the overall BCT intervention and not for each individual BCT.
Groups:
- Behavioral Change Techniques to Increase Walking: Individuals will receive daily text messages with the goal of increasing daily walking by 2,000 more steps five days per week. Participants will be enrolled for a baseline period lasting two weeks where their average daily activity level will be assessed using a Fitbit device to generate an average daily step counts. Following completion of baseline, participants will receive daily text messages of behavior change techniques (BCTs) for eight weeks. The four BCTs utilized in this study are: goal setting, action planning, self-monitoring of behavior, and feedback on behavior. Each BCT will be delivered to participants daily for a two-week block. Four blocks (one BCT per block) will be delivered to the participant. The order in which the BCT interventions are presented to participants will be randomized by the study statistician. The goal of the BCT text messages will be to encourage walking behavior.
  Behavioral Change Techniques: Four behavioral changes techniques (BCTs) will be administered to participants in random order.
Period: Baseline
Arm/Group | Behavioral Change Techniques to Increase Walking
Started | 72
Ineligible After Baseline | 11
Did Not Sign Addendum | 1
Completed | 60
Not Completed | 12
Period: Intervention
Arm/Group | Behavioral Change Techniques to Increase Walking
Started | 60
Completed | 59
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Change Techniques to Increase Walking
Number analyzed (Participants) | 60
Age, Customized [Count of Participants; unit: Participants]
  45 to 55 | 31
  56 to 65 | 27
  66 to 75 | 2
  Decline to Respond | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 48
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Within-person Change in Daily Steps.
Description: Participant steps will be assessed continuously using a Fitbit mobile device. Daily steps for participants will be aggregated by baseline and intervention phases to generate average daily steps in each phase. Changes in daily steps between baseline and intervention phases will be compared using Generalized Linear Mixed Model analyses. Changes in daily steps between intervention and baseline will be represented using a regression parameter.
Time Frame: Steps will be assessed continuously via worn activity tracker. Step counts will be aggregated and analyzed at the daily level. This will yield 70 daily measurements of physical activity over the course of the 10-week study.
Population: GLMM Regression for Change in Daily Steps Due to BCT Intervention
Measure: Number; unit: Daily Steps
Groups:
- Behavioral Change Techniques to Increase Walking: Individuals will receive daily text messages with the goal of increasing daily walking by 2,000 more steps five days per week. Following completion of baseline, participants will receive daily text messages of behavior change techniques (BCTs) for eight weeks. The four BCTs utilized in this study are: goal setting, action planning, self-monitoring of behavior, and feedback on behavior.
Arm/Group | Behavioral Change Techniques to Increase Walking
Number analyzed (Participants) | 60
Daily Steps
  Increase in Daily Steps Due to Intervention | 120.85
  Standard Error for Regression of Intervention on Daily Steps | 257.42

2. Primary Outcome: Participant Satisfaction With Personalized Trial Components.
Description: Participants will rate their satisfaction with the Personalized Trial overall and with individual elements of the trial in a satisfaction survey developed for this trial. Participants will rate 9 items assessing satisfaction with methods and process of the trial on a 4-point Likert scale with responses ranging from "0 - Not at all satisfied" to "3 - Very satisfied". Higher scores indicate greater levels of satisfaction. Means and standard deviations will be reported for each element of satisfaction.
Time Frame: Assessed once after completion of the study at 10 weeks.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Behavioral Change Techniques to Increase Walking
Number analyzed (Participants) | 59
Score on a scale
  The behavior change techniques (BCTs) assigned to you | 2.10 (0.92)
  The frequency that each BCT was delivered to you (daily) | 2.38 (0.81)
  Video explanations and demonstrations of study devices and procedures | 2.06 (1.00)
  Text messaging for delivery of study interventions (BCTs) | 2.42 (0.84)
  Text messaging for reminders (e.g. sync your Fitbit) | 2.59 (0.73)
  Text messaging for data collection (i.e. surveys) | 2.60 (0.70)
  Use of the fitbit device to track your activity and sleep | 2.71 (0.56)
  Study communications | 2.52 (0.73)
  Presentation of your results | 2.37 (0.88)

3. Secondary Outcome: Self-Efficacy for Walking
Description: This will be assessed using the Self-Efficacy for Walking (SE-W) scale,[1] an 10-item measure assessing patient's capabilities to walk for durations of 5 to 50 minutes. Items are scored from 0 to 100%, with scores of 0% indicating participants are "not at all confident" they could walk for that duration and scores of 100% indicating the participants are "highly confident" they could walk that duration. Items are average to create a total score, with higher scores indicating higher levels of beliefs about capabilities/self-efficacy.
Time Frame: Assessed at baseline, week 2, week 4, week 6, week 8, and week 10.
Reporting Status: Not Posted

4. Secondary Outcome: Participant Attitudes and Opinions Towards Personalized Trials.
Description: Participants will be asked via survey about their attitudes and opinions regarding the personalized trial implementation (e.g., Did the trial feel burdensome?). Participants will rate items on a 7-point Likert scale with responses ranging from "0 - Strongly Disagree" to "6 - Strongly Agree". Higher scores indicate greater levels of agreement. Scores on each item will be reported with means and standard deviations.
Time Frame: Assessed once after completion of the study at 10 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants are followed over 10 weeks (2 weeks of baseline and an 8-week intervention)
Arm/Group | Behavioral Change Techniques to Increase Walking
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04967313/Prot_SAP_000.pdf